CLINICAL TRIAL: NCT04205552
Title: Neoadjuvant Nivolumab Combination Treatment in Resectable Non-small Cell Lung Cancer Patients: Defining Optimal Combinations and Determinants of Immunological Response
Brief Title: Neoadjuvant Nivolumab Combination Treatment in Resectable Non-small Cell Lung Cancer Patients
Acronym: NEOpredict
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA224-063
Record Dates: First submitted 2019-12-16; First posted 2019-12-19 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: NSCLC Stage II; NSCLC, Stage IIIA; NSCLC, Stage I
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nivolumab (Experimental): Nivolumab 2 cycles, every two weeks (q2w)
  o Nivolumab 240 mg i.v. over 30 min
  Interventions: Drug: Nivolumab 10 MG/ML Intravenous Solution
- Nivolumab/Relatlimab (80 mg) (Experimental): Nivolumab/Relatlimab (80 mg) 2 cycles, every two weeks (q2w)
  * Nivolumab 240 mg i.v. over 30 min
  * Relatlimab 80 mg i.v. over 30 min (within 30 min of nivolumab)
  Interventions: Drug: Nivolumab 10 MG/ML Intravenous Solution; Drug: Relatlimab 10 MG/ML Intravenous Solution
- Nivolumab/Relatlimab (240 mg) (Experimental): Nivolumab/Relatlimab (240 mg) 2 cycles, every two weeks (q2w)
  * Nivolumab 240 mg i.v. over 30 min
  * Relatlimab 240 mg i.v. over 30 min (within 30 min of nivolumab)
  Interventions: Drug: Nivolumab 10 MG/ML Intravenous Solution; Drug: Relatlimab 10 MG/ML Intravenous Solution

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML Intravenous Solution — Neoadjuvant 2 cycles, every two weeks (q2w) Nivolumab 240 mg i.v. over 30 min
Drug: Relatlimab 10 MG/ML Intravenous Solution — Neoadjuvant 2 cycles, every two weeks (q2w) Relatlimab 80 mg i.v. over 30 min
  Arms: Nivolumab/Relatlimab (240 mg); Nivolumab/Relatlimab (80 mg)

SUMMARY:
The primary objective of this study is to determine the feasibility of four weeks of preoperative immunotherapy with Nivolumab, and Nivolumab plus Relatlimab in patients with early stage or locally advanced non-small cell lung cancer eligible for curative resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed non-small cell lung cancer (NSCLC) eligible for anatomic resection (Clinical stages I B, II and selected stage III A)
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Sufficient pulmonary function to undergo curative lung cancer surgery
* Adequate hematological, hepatic and renal function parameters:
* Sufficient cardiac left ventricular defined as left ventricular ejection fraction (LVEF) ≥ 50% documented either by echocardiography or multigated acquisition scan (MUGA)
* Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures

Exclusion Criteria:

* Active or history of autoimmune disease or immune deficiency
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration
* Subjects who have undergone organ transplant or allogeneic stem cell transplantation
* Uncontrolled or significant cardiovascular disease
* Patients with active neurological disease
* Active malignancy or a prior malignancy within the past 3 years
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study medication
* Peripheral polyneuropathy NCI CTCAE Grade ≥ 2
* History of gastric perforation or fistulae in past 6 months
* Serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment.
* The patient has undergone major surgery within 28 days prior to enrollment except staging mediastinoscopy, diagnostic Video Assisted Thoracoscopic Surgery (VATS) or implantation of a venous port-system.
* Any other concurrent preoperative antineoplastic treatment including irradiation
* Pregnant/Breastfeeding women
* Subjects with history of severe toxicity or life-threatening toxicity (grade 3 or 4) related to prior immune therapy
* Prior treatment with Lymphocyte-activation gene 3 (LAG-3) targeting Agent
* Previous treatment with Nivolumab or Relatlimab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of four weeks of preoperative immunotherapy with Nivolumab, Nivolumab plus Relatlimab (80 mg), and Nivolumab plus Relatlimab (240 mg) | Within 43 days after first study medication

SECONDARY OUTCOMES:
Estimation of pathological tumor response rate | Within 43 days after first study medication (day of surgery)
Estimation of curative (R0) resection rate | Within 43 days after first study medication (day of surgery)
Objective radiological response rate | After 3, 6, 9 and 12 months post-surgery
  Objective radiological response rate per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1
Disease-free survival rate at 12 months | 12 months
  Assessment of disease-free survival rate at 12 months per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1
Overall survival rate at 12 months | 12 months
Morbidity | within 90 days after surgery
  Estimation of morbidity within 90 days after surgery
Mortality | within 90 days after surgery
  Estimation of mortality within 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schuler, Prof. Dr., Principal Investigator — University Hospital, Essen
Locations (4):
- Jessa Hospital Hasselt, Hasselt, Belgium
- Germany (2):
  - University Hospital Essen, Essen
  - Thoraxklinik Heidelberg gGmbH-Universitätsklinikum Heidelberg, Heidelberg
- Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schuler M, Cuppens K, Plones T, Wiesweg M, Du Pont B, Hegedus B, Koster J, Mairinger F, Darwiche K, Paschen A, Maes B, Vanbockrijck M, Lahnemann D, Zhao F, Hautzel H, Theegarten D, Hartemink K, Reis H, Baas P, Schramm A, Aigner C. Neoadjuvant nivolumab with or without relatlimab in resectable non-small-cell lung cancer: a randomized phase 2 trial. Nat Med. 2024 Jun;30(6):1602-1611. doi: 10.1038/s41591-024-02965-0. Epub 2024 Apr 30. PMID 38689060
- See also: Neoadjuvant nivolumab with or without relatlimab in resectable non-small-cell lung cancer: a randomized phase 2 trial — https://pubmed.ncbi.nlm.nih.gov/38689060/